CLINICAL TRIAL: NCT07387172
Title: Relationships of B-cell Activating Factor Gene Polymorphisms With the Risk and Clinicopathological Features of Crohn's Disease.
Brief Title: Relationships of B-cell Activating Factor Gene Polymorphisms With Crohn's Disease.
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2026-01-201
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Extract whole genome DNA from peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CD patients: Patients diagnosed with Crohn's disease
- normal controls: gender- and age-matched normal controls

SUMMARY:
From January 2020 to December 2024, Crohn's disease(CD) patients and gender- and age-matched normal controls were collected from the Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. The aim of this research is to explore the associations of B-cell activating factor(BAFF) gene polymorphisms with the risk and clinicopathological characteristics of CD.

DETAILED DESCRIPTION:
From January 2020 to December 2024, a total of 310 CD patients and 514 gender- and age-matched normal controls were collected from the Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University.The genotypes of BAFF were determined by multiplex polymerase chain reaction-ligase detection reaction technique. Unconditional logistic regression was employed to analyze the distribution of BAFF gene polymorphisms between CD group and normal control group, as well as their influences on the clinicopathological characteristics of CD patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed CD based on comprehensive clinical, colonoscopy, histopathological, laboratory, and radiographic examination results

Exclusion Criteria:

* rheumatoid arthritis, systemic lupus erythematosus, intestinal tuberculosis, ischemic enteritis, radiation enteritis, tumors, etc

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There was no statistically significant difference in the gender ratio, average age, and proportion of smokers between CD group and normal control group. All study subjects are from the Zhejiang Han population who are not related by blood.
Sampling Method: Probability Sample
Enrollment: 824 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
the genotypes of BAFF | Baseline
  multiplex polymerase chain reaction-ligase detection reaction technique

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No